CLINICAL TRIAL: NCT00221390
Title: Randomized, Placebo-controlled, Double-blind Pilot Trial to Evaluate the Safety and Efficacy of Ropinirole in Motor Recovery After Stroke
Brief Title: Trial of Ropinirole in Motor Recovery After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS#2003-3096
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Cerebrovascular Accident; Hemiparesis
Keywords: stroke; Chronic stroke with hemiparesis
MeSH Terms: conditions — Stroke; Paresis | interventions — ropinirole; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ropinirole (+ physical therapy)
Drug: (vs.) Placebo + physical therapy

SUMMARY:
The purpose of this study is to assess efficacy, as well as safety, of Ropinirole in improving movement among patients with chronic stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability. Current treatments target injury and must be delivered within hours. A body of literature suggests that there are processes ongoing days-months after stroke that can be targeted therapeutically, and improve function. The current study evaluates one such potential therapy, the dopamine agonist ropinirole. The current study tests the hypothesis that patients with chronic stroke randomized to ropinirole+physiotherapy will show improved gait velocity over the 12 weeks of study participation as compared to patients randomized to placebo+physiotherapy. A secondary aim is to test the hypothesis that ropinirole will improve three secondary endpoints at 12 weeks after study entry: the proportion of patients with no significant disability (Barthel Index ≥ 95); overall motor status, measured with the arm/leg FM score; and overall physical function, defined as the score on the Stroke Impact Scale-16 (SIS-16). This study will also evaluate the safety of ropinirole in patients recovering from stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke onset 4 weeks-12 months prior
2. Stroke is radiologically confirmed as either (a) ischemic or (b) hemorrhagic
3. Minimum age 18
4. No significant pre-stroke disability
5. No other stroke in previous 3 months
6. Absence of major depression
7. Fugl-Meyer (FM) motor score of 23-83 out of 100
8. Functional Independence Measure (FIM) ambulation-subscore of 3 or more, and 50 foot walk takes longer than 15 seconds

Exclusion Criteria:

1. Significant daytime somnolence or any substantial decrease in alertness, language reception, or attention
2. Pregnant or lactating
3. Advanced liver, kidney, cardiac, or pulmonary disease
4. Orthostatic hypotension
5. Current use of ciprofloxacin, a centrally acting dopamine agonist, or a centrally active dopamine antagonist
6. A terminal medical diagnosis consistent with survival < 1 year
7. Coexistent major neurological disease
8. Coexistent major psychiatric disease
9. A history of significant alcohol or drug abuse in the prior 3 years
10. A coexistent disease characterized by an abnormality of CNS dopaminergic tone
11. Current enrollment in another investigational study related to stroke or stroke recovery
12. Contraindication to ropinirole prescription

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2003-10; Primary Completion 2007-02 (Actual); Study Completion 2007-05 (Actual)

SECONDARY OUTCOMES:
Barthel Index | Measured at weeks 1, 9, and 12
Leg motor Fugl-Meyer scale | Measured at baseline and weeks 1, 2, 4, 6, 7, 8, 9, and 12
Stroke Impact Scale-16 | Measured at weeks 1, 4, 7, 9, and 12
Gait endurance | Measured at weeks 1, 2, 4, 6, 7, 8, 9, and 12
Hamilton Depression Scale | Measured at baseline and weeks 1, 2, 9, and 12
Safety | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Cramer, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Background] Gresham GE, Duncan PW, Stason WB, Adams HP, Adelman AM, Alexander DN, Bishop DS, Diller L, Donaldson NE, Granger CV, Holland AL, Kelly-Hayes M, McDowell FH, Myers L, Phipps MA, Roth EJ, Siebens HC, Tarvin GA, Trombly CA. Post-Stroke Rehabilitation. Rockville, MD: U.S. Department of Health and Human Services. Public Health Service, Agency for Health Care Policy and Research, 1995.
- [Background] Rathore SS, Hinn AR, Cooper LS, Tyroler HA, Rosamond WD. Characterization of incident stroke signs and symptoms: findings from the atherosclerosis risk in communities study. Stroke. 2002 Nov;33(11):2718-21. doi: 10.1161/01.str.0000035286.87503.31. PMID 12411667
- [Background] Dobkin BH. Neurologic Rehabilitation. Philadelphia: FA Davis, 1996
- [Background] Nudo RJ. Recovery after damage to motor cortical areas. Curr Opin Neurobiol. 1999 Dec;9(6):740-7. doi: 10.1016/s0959-4388(99)00027-6. PMID 10607636
- [Background] Cramer SC, Chopp M. Recovery recapitulates ontogeny. Trends Neurosci. 2000 Jun;23(6):265-71. doi: 10.1016/s0166-2236(00)01562-9. PMID 10838596
- [Background] Finklestein S, Campbell A, Baldessarini RJ, Moya KL, Haber SN. Late changes in cerebral monoamine metabolism following focal ventrolateral cerebrocortical lesions in rats. Brain Res. 1985 Oct 7;344(2):205-10. doi: 10.1016/0006-8993(85)90796-6. PMID 2412650
- [Background] Finklestein S, Campbell A, Stoll AL, Baldessarini RJ, Stinus L, Paskevitch PA, Domesick VB. Changes in cortical and subcortical levels of monoamines and their metabolites following unilateral ventrolateral cortical lesions in the rat. Brain Res. 1983 Jul 25;271(2):279-88. doi: 10.1016/0006-8993(83)90290-1. PMID 6193832
- [Background] Boyeson MG, Feeney DM. Striatal dopamine after cortical injury. Exp Neurol. 1985 Aug;89(2):479-83. doi: 10.1016/0014-4886(85)90107-4. PMID 4018214
- [Background] Stroemer RP, Kent TA, Hulsebosch CE. Enhanced neocortical neural sprouting, synaptogenesis, and behavioral recovery with D-amphetamine therapy after neocortical infarction in rats. Stroke. 1998 Nov;29(11):2381-93; discussion 2393-5. doi: 10.1161/01.str.29.11.2381. PMID 9804653
- [Background] Cramer SC, Nelles G, Benson RR, Kaplan JD, Parker RA, Kwong KK, Kennedy DN, Finklestein SP, Rosen BR. A functional MRI study of subjects recovered from hemiparetic stroke. Stroke. 1997 Dec;28(12):2518-27. doi: 10.1161/01.str.28.12.2518. PMID 9412643
- [Background] Feeney DM, Gonzalez A, Law WA. Amphetamine, haloperidol, and experience interact to affect rate of recovery after motor cortex injury. Science. 1982 Aug 27;217(4562):855-7. doi: 10.1126/science.7100929.
- [Background] Gladstone DJ, Black SE. Enhancing recovery after stroke with noradrenergic pharmacotherapy: a new frontier? Can J Neurol Sci. 2000 May;27(2):97-105. PMID 10830340
- [Background] Goldstein LB. Potential impact of drugs on poststroke motor recovery. In: L. B. Goldstein, ed. Restorative Neurology. Advances in pharmacotherapy for recovery after stroke. Armonk, NY: Futura Publishing Co., 1998:241-256.
- [Background] Scheidtmann K, Fries W, Muller F, Koenig E. Effect of levodopa in combination with physiotherapy on functional motor recovery after stroke: a prospective, randomised, double-blind study. Lancet. 2001 Sep 8;358(9284):787-90. doi: 10.1016/S0140-6736(01)05966-9. PMID 11564483
- [Background] Sullivan KJ, Knowlton BJ, Dobkin BH. Step training with body weight support: effect of treadmill speed and practice paradigms on poststroke locomotor recovery. Arch Phys Med Rehabil. 2002 May;83(5):683-91. doi: 10.1053/apmr.2002.32488. PMID 11994808
- [Background] Richards C, Malouin F, Dumas F, Tardif D. Gait velocity as an outcome measure of locomotor recovery after stroke. In: C. R and O. C, eds. Gait Analysis: Theory and Application. St. Louis: Mosby, 1995:355-364.
- [Background] Potter JM, Evans AL, Duncan G. Gait speed and activities of daily living function in geriatric patients. Arch Phys Med Rehabil. 1995 Nov;76(11):997-9. doi: 10.1016/s0003-9993(95)81036-6. PMID 7487453
- [Background] Nieoullon A. Dopamine and the regulation of cognition and attention. Prog Neurobiol. 2002 May;67(1):53-83. doi: 10.1016/s0301-0082(02)00011-4. PMID 12126656
- [Background] Medico M, De Vivo S, Tomasello C, Grech M, Nicosia A, Castorina M, D'Agata MA, Rampello L, Lempereur L, Drago F. Behavioral and neurochemical effects of dopaminergic drugs in models of brain injury. Eur Neuropsychopharmacol. 2002 Jun;12(3):187-94. doi: 10.1016/s0924-977x(02)00010-x. PMID 12007669
- [Background] Bracha HS, Lyden PD, Khansarinia S. Delayed emergence of striatal dopaminergic hyperactivity after anterolateral ischemic cortical lesions in humans; evidence from turning behavior. Biol Psychiatry. 1989 Feb 1;25(3):265-74. doi: 10.1016/0006-3223(89)90174-1. PMID 2914151
- [Background] Nutt JG, Fellman JH. Pharmacokinetics of levodopa. Clin Neuropharmacol. 1984;7(1):35-49. doi: 10.1097/00002826-198403000-00002. No abstract available. PMID 6367973
- [Derived] Cramer SC, Dobkin BH, Noser EA, Rodriguez RW, Enney LA. Randomized, placebo-controlled, double-blind study of ropinirole in chronic stroke. Stroke. 2009 Sep;40(9):3034-8. doi: 10.1161/STROKEAHA.109.552075. Epub 2009 Jun 11. PMID 19520987